CLINICAL TRIAL: NCT04219839
Title: Duke Transplant University: A Digital Patient Education Portal
Brief Title: Duke Transplant University
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Haller Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO00102663
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2021-10

CONDITIONS: Kidney Transplant; Complications; Patient Empowerment; Medication Adherence; Patient Satisfaction
Keywords: patient education post-kidney transplant
MeSH Terms: conditions — Patient Participation; Medication Adherence; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 to either receive intervention (usual care + videos) or no intervention (usual care only.)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOC only patient education post- kidney transplant (No Intervention): Participants in this group will receive only SOC patient education following kidney transplant
- SOC + Videos for patient education post-kidney transplant (Experimental): Participants in this group receive SOC patient education following kidney transplant and access to educational videos designed specifically for post-kidney transplant patients.
  Interventions: Behavioral: SOC + Educational Videos Designed Especially for post-transplant patients

INTERVENTIONS:
Behavioral: SOC + Educational Videos Designed Especially for post-transplant patients — Patient focused videos (3-5 minutes each) with topics that will include: What to Expect After Transplant, What is the Kidney, Understanding your Labs, Transplant Medications, General Medical Care Post-Transplant, When to Call your Coordinator, and Self-Management/Sick Day protocols. Video curriculum will be offered in two ways. First, tablet computers with active links to each video will be available in kidney transplant clinic. At provider/coordinator discretion, study participants may also view videos while waiting for other appointments. In addition, for patients with smartphones who consent to this, a desktop link will be provided to the transplant video curriculum webpage (mobile friendly view).
  Arms: SOC + Videos for patient education post-kidney transplant

SUMMARY:
The purpose of this research study is to determine the effectiveness of educational videos for patients who have just had kidney transplant compared to usual patient education practices. Eligible patients will have the opportunity to enroll in this study after their transplant procedure either before hospital discharge or at their first follow up clinic visit.

DETAILED DESCRIPTION:
Participants will then complete a demographic survey and knowledge assesment to establish their baseline of knowledge regarding post-transplant care, medication adherence and patient satisfaction. Participants will then be randomly selected to receive either the usual patient education care provided for patients following kidney transplant, or to receive the usual care plus access to educational videos designed especially for post- transplant patients. Videos can be viewed on a tablet computer with their transplant team during clinic visits and at home using a smartphone.

At 3 months post-transplant, all participants will be asked to repeat the knowledge assessment. Hospital re-admissions and patient satisfaction will be measured at 6 months after transplant.

ELIGIBILITY:
Inclusion Criteria:

* recent kidney transplant recipients
* competent with the capacity to give legal written consent

Exclusion Criteria:

* Unable to sign informed consent.
* Patients with delirium, dementia, or other cognitive impairment that would not allow informed consent to enter the study.
* patients with severe vision or auditory impairment who are unable to view or hear electronic videos at close range.
* patients who are unable to understand the English language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Change in patient transplant knowledge during intervention as measured by the scores from the "Transplant Knowledge" block within the Duke Transplant University Assessment | Baseline to 3 months
  Change will be measured by comparing the scores from the Transplant Knowledge assessments completed at baseline and 3 months.
Change in perceptions of self-efficacy as measured by the scores from the "Self-Efficacy and Resiliency" assessment within the Duke Transplant University Assessment | Baseline to 3 months
  Change will be measured by comparing the scores from the Self-Efficacy and Resiliency assessments completed at baseline and 3 months.
Number of medication errors made post-transplant as measured by pillbox errors | 1 month, 2 months and 3 months
  The number of medication errors will be measured by counting number of pill box errors identified by pharmacist's review of patient's pillbox during transplant follow up clinic visits conducted at 1 month, 2 months and 3 months.

SECONDARY OUTCOMES:
Patients' satisfaction with the transplant experience as measured by satisfaction ratings | Baseline and 6 months
  Patients' satisfaction with the transplant experience will be measured by the rating scores from "general satisfaction" metrics.
Number of hospital re-admissions post transplant | Baseline to 6 months
  Hospital re-admissions will be collected from patient report and review of electronic medical record

CONTACTS AND LOCATIONS:
Overall Officials: John K Roberts, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No